CLINICAL TRIAL: NCT02676336
Title: A Randomized Double-blind, Placebo Controlled, Multi-center Study to Evaluate the Safety, Tolerability and Potential Effects of the Dietary Supplement Violet™ Molecular Iodine (I2) on Breast Health in Women With Cyclic Breast Discomfort and Tenderness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16VBHB
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Fibrocystic Breast Condition (FBC)
Keywords: FBC; cyclic mastalgia; breast discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Violet™ Iodine (Active Comparator): 3mg molecular iodine (I2) daily
  Interventions: Dietary Supplement: Violet™ Molecular Iodine (I2)
- Placebo (Placebo Comparator): 3mg placebo daily
  Interventions: Other: Placebo
- Cross-over (Active Comparator): Subjects on placebo will be offered 3 months of active post-treatment
  Interventions: Dietary Supplement: Violet™ Molecular Iodine (I2)

INTERVENTIONS:
Dietary Supplement: Violet™ Molecular Iodine (I2)
  Arms: Cross-over; Violet™ Iodine
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, multi-center study to evaluate the safety, tolerability and potential effects of dietary supplement Violet™ Iodine on breast health in women with cyclic breast discomfort and tenderness to eliminate the evaluation of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy premenopausal females ≥ 18 years of age
* BMI 20.0 - 29.9 kg/m2 (± 1 kg/m2)
* Females of childbearing potential must agree to use a reliable and consistent method of birth control in the Investigator's opinion, excluding depot contraceptives and Explanon, and have a negative urine pregnancy test result. Hormonal contraceptives such as oral contraceptives, birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing) are all acceptable as long as the subject is on a stable dose and agrees not to change during the study period
* No apparent health conditions that in the investigator's opinion would interfere with study participation, compliance or interpretation of endpoints or would not be in the best interest of the subject
* Moderate to severe cyclic breast discomfort of at least 4 days per month (discomfort ≥4 on a 0-10 scale)
* No known medical or psychological condition that in the investigator's opinion could interfere with study participation
* Agrees to comply with all study related procedures and visits including access to a smartphone (Android or iOS) and ability to enter daily diary information via a smart phone app
* Capable of reading and understanding study related materials (in English or French) and has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
* Perimenopausal or irregular menstrual cycles
* Women who have had an oophorectomy
* Known thyroid condition or currently taking any thyroid medications
* Prior bariatric surgery or other interventions or medications that might affect gastric pH
* Use of iodine supplementation, Tamoxifen, Lupron, or Danazol, in the last 6 months
* Clinically significant abnormal laboratory results at Screening
* Breast implant surgeries that have not fully healed or have ongoing problems associated with the implant (i.e. seroma, infection etc.)
* Planned elective surgeries to occur during participation in the study
* Known allergy or sensitivity to study product ingredients (e.g. Iodine)
* History of alcohol or drug abuse within the past year
* Use of medicinal marijuana within the past year
* Participation in a clinical research trial within 30 days prior to randomization or plans to participate in any other study during the next 11 months
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures, may confound interpretation of study outcome measures (such as another condition) or which may pose significant risk to the subject

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in self assessed cyclic breast discomfort | After 6 months of active treatment with molecular iodine (I2) compared to placebo

CONTACTS AND LOCATIONS:
Locations (2):
- KGK Synergize, Orlando, Florida, United States
- KGK Synergize, London, Ontario, Canada